CLINICAL TRIAL: NCT00330876
Title: Open-Label, Long-Term (> 1 Year) Extension Study of Pitavastatin in Elderly Patients With Primary Hypercholesterolemia or Combined Dyslipidemia
Brief Title: Study of Pitavastatin in Elderly Patients With Primary Hypercholesterolemia or Combined Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Neil Hounslow, Kowa Research Europe
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-104-308EU
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Hypercholesterolemia; Dyslipidemias
Keywords: pitavastatin; hypercholesterolemia; combined dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin 2 mg QD (Experimental): Pitavastatin 2 mg once daily
  Interventions: Drug: Pitavastatin
- Pitavastatin 4 mg QD (Experimental): Pitavastatin 4 mg once daily
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Pitavastatin

SUMMARY:
This is an open-label extension study of NK-104-306 (NCT00257686) for elderly patients with hypercholesterolemia or combined dyslipidemia.

DETAILED DESCRIPTION:
This was an open-label study of 60 weeks duration in elderly patients (≥65 years) with primary hypercholesterolemia or combined dyslipidemia who completed the 12 week treatment in study NK-104-306 and who met the inclusion/exclusion criteria. Patients who qualified started open-label treatment with pitavastatin 2 mg QD. The dose of pitavastatin could be increased to 4 mg QD after at least 8 weeks of treatment at 2 mg QD, in patients who failed to attain their LDL-C target.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 65 years of age
* Primary hypercholesterolemia
* Combined dyslipidemia
* Completed study NK-104-306 (NCT00257686)

Exclusion Criteria:

* Failed to complete study NK-104-306(NCT00257686)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 545 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, MD, Study Director — Medical Director
Locations (59):
- Denmark (3):
  - Copenhagen University Hospital, Copenhagen
  - Medical Center, Copenhagen
  - CCBR A/S, Vejle
- Germany (17):
  - Kardiologische Gemeinschaftspraxis Prof. Reifart, Bad Soden/Taunus
  - Praxis Dr. Boenninghoff, Beckum
  - Klinische Forschung Berlin Mitte, Berlin
  - GWT-TUK GmbH, Zentrum fur Klinische Studien, Dresden
  - Gemeinschaftspraxis Dr. Krause, Th. Menke, Goch
  - Klinische Forschung Hamburg, Hamburg
  - Innere Medizin I/Medizinische Klinik, Heidelberg
  - Gemeinschaftspraxis H. Holz Dr. Med, K. W. Klingl, Lampertheim
  - ZET-Studien GmbH Leipzig, Leipzig
  - Internistische Gemeinschaftspraxis, Mainz
  - Praxis Dr. Wachter, Mannheim
  - Gemeinschaftspraxis Melcherstaette, Melcherstaette
  - Gemeinschaftspraxis Dr. Senftleber, Dr. Kohler, Messkirch
  - Praxisgemeinschaft im Kleinen Biergrund, Offenbach/M
  - Gemeinschaftspraxis Drs. Mockesch, Weinheim
  - Intermed Institud Fur Klinische Forschung und Arzn, Wiesbaden
  - Gemeinschaftspraxis Dr. Emden, Frank Drewes, Worpswede
- Israel (9):
  - Department of Internal Medicine, Soroka Medical Center, Beersheva
  - Department of Internal Medicine A, Rambal Medical Center, Haifa
  - Department of Internal Medicine, Wolfson Medical Center, Holon
  - Center for Research, Hadassah University Hospital, Jerusalem Ein Kerem
  - Meir Hospital, Kfar Saba
  - Department of Medicine, Hadassah Medical Center, Mount Scopus Jerusalem
  - Department of Internal Medicine, Rivka Sieff Medical Center, Safed
  - Institute of Metabolic Diseases, Tel Aviv
  - Institute of Lipid & Atherosclerosis Research, Tel Litwinsky
- Netherlands (10):
  - Andromed Breda, Breda
  - Andromed Noord, Groningen
  - Vasculair Onderzoek Centrum Hoorn, Hoorn
  - Andromed Leiden, Leiden
  - Andromed Nijmegen, Nijmegen
  - Andromed Rotterdam, Rotterdam
  - Albert Schweitzer Ziekenhuis, Sliedrecht
  - Rivierenland Tiel, Tiel
  - Andromed Oost, Velp
  - Andromed Zoetermeer, Zoetermeer
- United Kingdom (20):
  - Oldfield Surgery, Bath
  - St James's Surgery, Bath
  - The Pulteney Practice, Bath
  - Birmingham Clinical Research Centre, Birmingham
  - Stonehill Medical Center, Bolton
  - Chorley Clinical Research Centre, Chorley
  - Saltash Health Center, Cornwall
  - Gomersal Lane Surgery, Dronfield
  - Townhead Research, Irvine
  - Crosby Clinical Research Centre, Liverpool
  - The Symons Medical Center, Maidenhead
  - Manchester Clinical Research Centre, Manchester
  - Greenwood Medical Center, Nottingham
  - Reading Clinical Research Centre, Reading
  - Elm Lane Surgery, Sheffield
  - Brook Lane Surgery, Southampton
  - Bradford Road Medical Center, Wiltshire
  - Rowden Medical Partnership, Wiltshire
  - The Porch Surgery, Wiltshire
  - The Burns Medical Practice, Yorkshire

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pitavastatin 2 mg QD | Pitavastatin 4 mg QD
Started | 449 | 90
Completed | 378 | 77
Not Completed | 71 | 13

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: Subjects who received at least one dose of Pitavastatin 2 or 4 mg once daily
Arm/Group | Safety Population
Number analyzed (Participants) | 539
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 539
Age Continuous [Mean (Standard Deviation); unit: years] | 70.3 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294
  Male | 245

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in LDL-C
Description: percent change from baseline in low density lipoprotein-cholesterol (LDL-C)
Time Frame: Baseline to 60 weeks
Population: Subjects with measurement at Week 60
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 2 mg QD | Pitavastatin 4 mg QD
Number analyzed (Participants) | 376 | 77
percent change | -43.18 (10.065) | -44.26 (10.764)

2. Secondary Outcome: Change From Baseline in Total Cholesterol
Description: Percent change from baseline in total cholesterol (TC)
Time Frame: Baseline to 60 weeks
Population: Subjects with a measurement at Week 60
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 2 mg QD | Pitavastatin 4 mg QD
Number analyzed (Participants) | 378 | 77
percent change | -28.27 (8.214) | -30.54 (8.226)

ADVERSE EVENTS:
Arm/Group | Pitavastatin 2 mg QD | Pitavastatin 4 mg QD
Serious Adverse Events (participants affected / at risk) | 51/449 | 7/90
Other Adverse Events (participants affected / at risk) | 286 | 24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 2 mg QD (N=449) | Pitavastatin 4 mg QD (N=90)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute mycocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cporonary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
hypoacusis (Ear and labyrinth disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Urethral stricture (Renal and urinary disorders) | 1 | 0
Daiphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pitavastatin 2 mg QD | Pitavastatin 4 mg QD
Nasopharyngitis (Infections and infestations) | 71/539 | 2/95
Urinary tract infection (Infections and infestations) | 26/539 | 4/95
Cystitis (Infections and infestations) | 26/539 | 1/95
Myalgia (Musculoskeletal and connective tissue disorders) | 44/539 | 4/95
Arthralgia (Musculoskeletal and connective tissue disorders) | 34/539 | 3/95
Osteaoarthritis (Musculoskeletal and connective tissue disorders) | 24/539 | 5/95
Cough (Respiratory, thoracic and mediastinal disorders) | 26/539 | 1/95
Hypertension (Vascular disorders) | 35/539 | 4/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days